CLINICAL TRIAL: NCT05405647
Title: Extra Corporeal Shock Wave Versus Kinesio Tape in the Treatment of Carpal Tunnel Syndrome for Post Menopausal Women
Brief Title: Extra Corporeal Shock Wave Versus Kinesio Tape in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Ebrahim El Refaye, assistant professor department of Physical Therapy for Women's Health, Faculty of Physical therapy, Cairo University, Egypt, Woman's Health University Hospital, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cairo Un115
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Carpal Tunnel Syndrome
Keywords: shock wave; kinesio tape; carpal tunnel syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Extracorporeal Shockwave Therapy; Athletic Tape

STUDY DESIGN:
Intervention Model Description: Fifty menopausal women with mild to moderate CTS will be selected randomly from outpatient clinic of the physical therapy department of El khazendara general hospital, Shobra to participate in this study,Group A: Represented the study group, it consisted of 25 patients who received a program of 6 session of Shock wave Therapy on the affected wrist,5 minute per session. Group B: Represented the control group, it consisted of 25 patients who received a program of kinesio tape application on the affected wrist for 3 days .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- shock wave therapy (Experimental): received a program of 6 session of Shock wave Therapy on the affected wrist,5 minute per session, and a frequency of 5 Hz., 1 sessions per week for 6 weeks.
  Interventions: Device: Shock wave Therapy; Device: kinesio tape
- kinesio tape (Experimental): kinesio tape application on the affected wrist for 3 days and then one day off and then another 3 days each week for 6 weeks.
  Interventions: Device: Shock wave Therapy; Device: kinesio tape

INTERVENTIONS:
Device: Shock wave Therapy — a program of 6 session of Shock wave Therapy on the affected wrist,5 minute per session and a frequency of 5 Hz., 1 sessions per week for 6 weeks.
Device: kinesio tape — kinesio tape application on the affected wrist for 3 days and then one day off and then another 3 days each week for 6weeks.

SUMMARY:
This study would be conducted to answer the following question: was there any difference between the effects of Shock wave versus Kinesio Tape in the treatment of carpal tunnel syndrome for post-menopausal women.

DETAILED DESCRIPTION:
Fifty menopausal women with mild to moderate CTS were selected randomly from outpatient clinic of the physical therapy department of El khazendara general hospital, Age was ranged from 45 - 55 years old.

Group A, consisted of 25 patients who received a program of 6 session of Shock wave Therapy on the affected wrist,5 minute per session. Group B Represented the control group, it consisted of 25 patients who received a program of kinesio tape application on the affected wrist for 3 days.

ELIGIBILITY:
Inclusion Criteria:

* -Age was ranged from 45 - 55 years old
* All subjects would not take analgesics by another route during the study.

Exclusion Criteria:

* Patients had previous carpal tunnel release.
* Skin over sensitivity of some patients to the tape.

Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-01-29 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Computerized electromyography | 6 weeks
  2 channel version with EMG/NCV/EP system, It was used to measure median motor distal latency (MMDL) before treatment and after 6 weeks of treatment for all patients

SECONDARY OUTCOMES:
Boston carpal tunnel questionnaire | 6 weeks
  The overall score for the functional-status scale was the mean of the ratings on the 8 daily activities. In this study BCTQ was translated and filled by the therapist

CONTACTS AND LOCATIONS:
Locations (1):
- Ghada Ebrahim Elrefaye, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No